CLINICAL TRIAL: NCT06042400
Title: Pilot Trial of Written Exposure Intervention for Metastatic Cancer Patients: The EASE Study
Brief Title: Trial of Written Exposure for Metastatic Cancer Patients (EASE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Joanna Arch, Associate Professor, University of Colorado, Boulder
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-0243
Record Dates: First submitted 2022-05-16; First posted 2023-09-18 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Cancer; Solid Tumor Cancer; Lymphoproliferative Disorders; Anxiety; Post-traumatic Stress Symptoms; Fear of Cancer Progression
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoproliferative Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single-arm pilot trial: all participants will receive intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EASE Written Exposure Intervention (Experimental): Assigned Intervention
  Interventions: Behavioral: Written Exposure Therapy

INTERVENTIONS:
Behavioral: Written Exposure Therapy — An innovative written exposure therapy intervention that addresses psychosocial needs commonly experienced by patients with late stage cancers.

SUMMARY:
In the face of imminent loss, many adults with metastatic cancer report a range of mental health challenges, including cancer-related trauma symptoms, fear of cancer progression and dying/death, anxiety, depression, and hopelessness, as well as physical symptoms such as fatigue and pain. Cancer patients may report feeling upset or haunted by imagined scenarios in a way that causes them distress and lowers their quality of life.

This study aims to look at the acceptability and feasability of a writing-based intervention for adults with late-stage or recurrent cancer, or actively treated blood cancer. The EASE study uses a writing-based approach to address an individual's worst-case scenario about cancer because previous studies have shown that similar approaches have shown promise in reducing fear in early-stage cancer survivors and among adults with PTSD (posttraumatic stress disorder). The EASE study represents a novel adaptation of this foundational work on written exposure therapy (WET) to address worst-case scenarios among adults with late stage cancers.

The EASE study will include 5 weekly one-on-one online video sessions with a trained therapist where participants will be coached through writing exercises based on a worst-case scenario related to their cancer experience.

DETAILED DESCRIPTION:
This single-arm pilot trial aims to look at the acceptability and feasibility of a writing-based intervention for adults with metastatic or recurrent cancer, or actively treated blood cancer.

The EASE intervention represents a novel adaptation of foundational work on written exposure therapy (WET) to address worst-case scenarios among adults with metastatic cancer, including cancer diagnosed at Stage III or IV, cancer that has recurred, or actively treated lymphoproliferative cancer. The study will consist of 5 weekly one-on-one online sessions with a trained graduate student therapist who will explain the approach and coach participants through writing exercises based on a worst-case scenario related to their fears about cancer.

Remote Delivery.

The intervention will be delivered remotely via videoconferencing software or videoconferencing plus phone. Phone sessions will be available as a backup if a participant has significant technical difficulties with Zoom. All sessions will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. English-speaking (able to speak, read, and write well in English)
3. Diagnosed with solid tumor cancer at Stage III (locally metastatic) or Stage IV (distantly metastatic) or solid tumor cancer that has recurred, or actively treated lymphoproliferative cancer (e.g., non-solid tumor cancer)
4. Report elevated cancer-related trauma symptoms or fear of cancer progression on the screening measures: IES-R, FoP-Q 12-item short version.
5. No moderate to severe dementia reported by patient or seen during eligibility confirmation in the medical chart
6. Are capable at time of consent of understanding and voluntarily consenting themselves to the study, attending EASE sessions, and completing the online sessions at home, confirmed by an Eastern Cooperative Group Performance Status Scale of 0 to 2. Given that the study does not require individuals to leave their home, we will make an exception for individuals endorsing an Eastern Cooperative Group Performance Status Scale score of 3 (confined to bed or chair for <50% of waking hours, able to do only limited selfcare) if they meet all other study criteria, including criteria 7.
7. Report that they are able and willing to complete all study procedures, including the online assessments and the intervention itself, including being physically able to write by hand or type for 30 minutes at a time and do weekly hour-long EASE sessions by Zoom.
8. Has access to a computer with internet connection or are willing to use a study-loaned computer tablet for the study duration, and are willing to conduct sessions via videoconferencing on a computer

Exclusion Criteria:

1. Current moderate or high suicide risk evaluated by the Columbia Suicide Severity Rating Scale (CSSRS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Cancer-related trauma symptoms | Assessed seven times: prior to the intervention (Pre), before each intervention session, 3 weeks after the intervention begins (Mid), 6 weeks after baseline (Post), at 1.5 and 3-month follow-up (FU)
  A primary outcome will be change in cancer-related trauma symptoms, assessed by the 22-item Impact of Events Scale-Revised. Possible scores range 0-88 with higher scores indicating greater distress/bother.
Fear of cancer progression | Assessed: prior to the intervention (Pre), before each intervention session, 3 weeks after the intervention begins (Mid), 6 weeks after baseline (Post), at 1.5 and 3-month follow-up (FU)
  A primary outcome will be change in fear of cancer progression, assessed by the 12-item Fear of Progression Questionnaire - Short Form and by the four general scale items from the Concerns about Recurrence Scale, with wording adapted to focus on cancer progression rather than recurrence. Range: 12-60, higher scores are associated with higher fear of cancer progression.
Intervention acceptability | Assessed in order to compare values at 2 timepoints: 6 weeks after baseline (Post) and separately at 1.5-month follow-up (FU)
  Assessed with the Acceptability of Intervention Scale. Possible scores range from 4-20, with higher scores indicating greater intervention acceptability.
Intervention Feasibility | Assessed at each intervention session 1-5, 1 to 5 weeks after baseline.
  For participants who begin the intervention, at least 70% complete all intervention sessions

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-8) | Assessed: prior to the intervention (Pre), 3 weeks after the intervention begins (Mid), 6 weeks after baseline (Post),, at 1.5 and 3-month follow-up (FU)
  Patient-reported depression symptom questionnaire. Range is 0 to 24. Higher scores indicate more depression symptoms
Generalized Anxiety Disorder-7 Questionnaire | Assessed: prior to the intervention (Pre), 3 weeks after the intervention begins (Mid), 6 weeks after baseline (Post), at 1.5 and 3-month follow-up (FU)
  Patient-reported anxiety symptom questionnaire. Possible scores range from 0-21, with higher scores indicating more anxiety symptoms
The Death Attitude Profile-Revised, Fear of Death and Death Avoidance Scales | Assessed: prior to the intervention (Pre), 3 weeks after the intervention begins (Mid), 6 weeks after baseline (Post), at 1.5 and 3-month follow-up (FU)
  Patient-reported fear of death and dying questionnaire. Possible scores range from 12-84, with higher scores indicating greater fear of death and dying
Hopelessness Assessment in Illness Questionnaire 8-item | Assessed: prior to the intervention (Pre), 3 weeks after the intervention begins (Mid), 6 weeks after baseline (Post), at 1.5 and 3-month follow-up (FU)
  Patient-reported hopelessness specifically intended for use with adults with incurable cancer. Possible scores range 0-16, with higher scores indicating greater hopelessness.
The Patient Reported Outcome Measurement Information System (PROMIS) Fatigue-Short Form v1.0 | Assessed: prior to the intervention (Pre), 3 weeks after the intervention begins (Mid), 6 weeks after baseline (Post), at 1.5 and 3-month follow-up (FU)
  Patient-reported levels of fatigue. Possible scores range 6-30, with higher scores indicating greater fatigue.
The Patient Reported Outcome Measurement Information System (PROMIS) Pain Interference-Short Form v1.0 | Assessed: prior to the intervention (Pre), 3 weeks after the intervention begins (Mid), 6 weeks after baseline (Post), at 1.5 and 3-month follow-up (FU)
  Patient-reported dimension of pain interference (e.g., the extent to which pain interferes with daily life and life roles). Possible scores range 6-30, with higher scores indicating greater pain.
Emotional Approach Coping Scale (COPE): Avoidance coping (process measure) | Assessed: prior to the intervention (Pre), 3 weeks after the intervention begins (Mid), 6 weeks after baseline (Post), at 1.5 and 3-month follow-up (FU)
  Patient-reported coping through avoidance using three avoidance coping scales (mental disengagement, denial, physical disengagement) with cancer as the anchor. Possible scores range 8-28, with higher scores indicating greater denial, mental and behavioral disengagement.
Five Factor Mindfulness Questionnaire, Nonjudge and nonreact scales (process measure) | Assessed: prior to the intervention (Pre), 3 weeks after the intervention begins (Mid), 6 weeks after baseline (Post), at 1.5 and 3-month follow-up (FU)
  Patient-reported coping through acceptance. Possible scores range 15-75, with higher scores reflecting greater nonreactivity and nonjudging of inner experience.
Valuing Questionnaire | Assessed: prior to the intervention (Pre), 3 weeks after the intervention begins (Mid), 6 weeks after baseline (Post), at 1.5 and 3-month follow-up (FU)
  Valued engagement in daily life. Possible scores range 0-30 for each of the two subscales with higher scores indicating greater engagement and sense of purpose in life.
Self-compassion Scale-Short Form | Assessed: prior to the intervention (Pre), 3 weeks after the intervention begins (Mid), 6 weeks after baseline (Post), at 1.5 and 3-month follow-up (FU)
  Self-compassion questionnaire. Possible scores range 12-60 with higher scores indicating higher self-compassion.

OTHER OUTCOMES:
Intervention Acceptability: Session Feedback Questionnaire | Once weekly during intervention period from Pre to Post (6 weeks after baseline, e.g., at the end of each weekly session during the intervention period)
  Participant value of the session will be assessed through the Session Feedback. Possible scores range 4-20, with higher scores indicating higher value and acceptability of the session.
Intervention Acceptability: Client Satisfaction Questionnaire-8 | Assessed and reported two times: 6 weeks after baseline (Post), 3-month follow-up (FU)
  Participant satisfaction will be measured using the Client Satisfaction Questionnaire-8 (adapted to the current intervention). Possible scores range 8-32, with higher scores indicating more satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Arch, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No